CLINICAL TRIAL: NCT04372524
Title: Biomarker Verification in Pediatric Chronic Graft-Versus-Host Disease: Applied Biomarkers to Minimize Long Term Effects of Childhood/Adolescent Cancer Treatment (ABLE) / Pediatric Transplantation & Cellular Therapy Consortium (PTCTC)
Brief Title: Biomarker Verification in Pediatric Chronic GvHD: ABLE 2.0 / PTCTC GVH 1901 Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kirk Schultz, Professor of Pediatrics, University of British Columbia
Other Study IDs: H19-02032
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Chronic Graft-versus-Host-Disease; Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation; Blood Cancer; Non-Malignant Hematologic and Lymphocytic Disorder
Keywords: cGvHD; HSCT; L-aGvHD; Biomarkers; Blood; Pediatric; Adolescent; Chronic Graft-versus-Host-Disease; Hematopoietic Stem Cell Transplant; Late acute Graft-versus-Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic HSC Transplant recipients: Five possible patient scenarios are anticipated to occur in those who underwent allogeneic HSCT:
  * Early event (e.g. death, non-engraftment) occurring before day 100.
  * No late-acute or chronic GvHD ever develops at any time point in the first year post-transplant (regardless of whether or not classical acute GvHD develops in the first 100 days after transplant).
  * Early-onset chronic GvHD (including overlap syndrome) occurred before day 60.
  * Early-onset chronic GvHD (including overlap syndrome) occurred between day 60 and day 100.
  * Chronic GvHD after Day 100, Late-acute GvHD (de-novo or recurrent) after day 100, or cases of overlap syndrome occurred after day 100.

SUMMARY:
This study will validate a previously developed pediatric prognostic biomarker algorithm aimed at improving prediction of risk for the later development of chronic graft-versus-host disease (cGvHD) in children and young adults undergoing allogeneic hematopoietic stem cell transplant.

By developing an early risk stratification of patients into low-, intermediate-, and high-risk for future cGvHD development (based upon their biomarker profile, before the onset of cGvHD), pre-emptive therapies aimed at preventing the onset of cGvHD can be developed based upon an individual's biological risk profile.

This study will also continue research into diagnostic biomarkers of cGvHD, and begin work into biomarker models that predict clinical response to cGvHD therapies.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (cGvHD) occurs when the new donor immune system "attacks" tissues in the recipient following allogeneic hematopoietic stem cell transplantation (HSCT), leading to chronic inflammation, scarring and fibrosis, impaired immunity (including immune deficiency and immune dysregulation), and altered organ system functioning. Almost any organ or system has the potential to be affected by cGvHD, although eight organ systems are classically involved, including the skin, eyes, mouth, lungs, liver, gastrointestinal tract, genitourinary tract, and the musculoskeletal system.

The investigators will be enrolling allogeneic HSCT recipients before conditioning, following these patients prospectively until 12-months (+/- 1 month) post-transplant for the development of all forms of GvHD (classical acute, late acute and chronic GvHD), collecting blood samples at day +60 (+/- 7 days), day +100 (+/- 14 days), and at the onset of either late acute or chronic GvHD. Two extra blood samples will be collected exclusively from HAPLO transplant recipients, who never developed any late-acute GvHD or chronic GVHD at the 6- and 12-month post-transplant time points. In addition, clinical data will be collected at different time points.

Case report forms of standard transplant related data will be completed and entered into a REDCap database.

Blood samples will be drawn and shipped to the Central Laboratory in Vancouver, BC, Canada, processed, analyzed, and the final biomarker risk algorithm completed. Selected clinicians will be offered to complete a short survey asking about their perception of the feasibility of altering their approach to cGvHD management based upon these results.

If chronic GvHD develops at any time after transplant (day 0 to 1 year), or if any form of GvHD occurs at or after day +100 (whether late acute, chronic GvHD, or overlap syndrome), a blood sample will be drawn before escalating immune suppression, and the onset GvHD case report form will be completed following the protocol. If chronic GvHD is confirmed, an additional CRF will be submitted at 24-months (+/- 3 months) post-transplant to document new chronic GvHD manifestations, severity, and response to therapy.

Study participants will have between 2 and 4 blood samples drawn over the course of 1-year post-transplant, depending upon their event and GvHD status.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Any indication for allogeneic hematopoietic stem cell transplant (malignant or non-malignant)
2. Age 0 - 24.99 years at the time of transplant (on day 0)
3. Any conditioning regimen (including myeloablative or reduced-toxicity/reduced-intensity)
4. Any graft source (bone marrow, peripheral blood, cord blood)
5. Any graft-versus-host disease prophylaxis strategy, including serotherapy such as ATG or alemtuzumab
6. Haploidentical transplants, including post-transplant cyclophosphamide and alpha-beta TCR depletion, are allowed

EXCLUSION CRITERIA:

1. Second or greater allogeneic transplant
2. Weight 7 kg or less
3. Pure CD34+ selected haploidentical stem cell transplant (not including CD34 enrichment used in alpha-beta TCR depleted haploidentical transplants, which is allowed)
4. Inability of a center to follow a patient for the development of late-acute and chronic GVHD until 1-year post-transplant (referral sites who transplant patients from outside institutions should not enroll participants if sending back to the referring site early, such that long-term follow up, blood, and data collection cannot be assured).

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and adult (under age of 25 y.o.) patients undergoing allogeneic HSCT (hematopoietic stem cell transplantation) before the start of the conditioning regimen.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Day 60 blood sample collection | Day 60 (+/- 7 days) post-transplant
  Validation of prognostic and diagnostic power of cGvHD biomarkers and testing of the biomarker assay performance of Day 60 post-transplant blood sample. Using this algorithm-based assay the investigators will attempt to develop risk assignment for cGvHD and L-aGvHD at Day 60 and determine whether this time point has a similar (or improved) predictive value to the day +100 (+/-14 days). Flow Cytometry and ELISA assays will be used for biomarker measurement.
Day 100 blood sample collection | Day 100 (+/- 14 days) post-transplant
  Validation of prognostic and diagnostic power of cGvHD biomarkers and testing of the biomarker assay performance of Day 100 post-transplant blood sample (diagnostic biomarkers). Using this algorithm-based assay the investigators will attempt to develop risk assignment for cGvHD and L-aGvHD at Day 100. Flow Cytometry and ELISA assays will be used for biomarker measurement.
Onset CvHD blood sample collection | The day of initial diagnosis
  Validation of prognostic and diagnostic power of cGvHD biomarkers and testing of the biomarker assay performance of the GvHD onset blood sample. The investigators will attempt to determine whether biomarkers present at the onset of new late-acte GvHD developing after day +100 (diagnostic biomarkers) or are similar to or different than at the onset of chronic GvHD. Flow Cytometry and ELISA assays will be used for biomarker measurement.
Baseline transplant clinical data collection at Day 0 | Between day 0 (day of transplant) and day +21
  Baseline Transplant Data Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at Day 60 | Day 60 (+/- 7 days) post-transplant
  Day 60 Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at Day 100 | Day 100 (+/- 14 days) post-transplant
  Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at 6 months | 6 Months (+/- 1 month) post-transplant
  Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at 12 months | 12 Months (+/- 1 month) post-transplant
  Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at 24 months | 24 Months (+/- 1 month) post-transplant
  Case Report Form to be completed. Clinical data will be used in data analysis.
Clinical data collection at onset of GvHD | At the time of diagnosis
  Case Report Form to be completed. Clinical data will be used in data analysis.

SECONDARY OUTCOMES:
Demonstration of identifiable and reproducible differences in diagnostics of cGvHD and L-aGvHD | At the end of the study by year 2025
  Metrics to measure this outcome will employ the difference in biomarkers (in combination with clinical manifestation) that can be used to discriminate between cGvHD and L-aGvHD and aid clinicians in establishing a more accurate diagnosis. Laboratory procedure and statistical data analysis will be used to achieve this.
Determination of patient's risk profile and prediction of treatment responses | At the end of the study by year 2025
  Utilizing cGvHD specific biomarkers, clinicians will be able to predict patient's treatment responses and chose the more accurate and effective treatment options.

OTHER OUTCOMES:
6 Month HAPLO blood sample collection | 6 Months (+/- 1 month) post-transplant
  Blood sample from haploidentical transplant recipients who did not develop late-acute or chronic GvHD
12 Month HAPLO blood sample collection | 12 Months (+/- 1 month) post-transplant
  Blood sample from haploidentical transplant recipients who did not develop late-acute or chronic

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Schultz, MD, Principal Investigator — University of British Columbia / BC Children's Hospital Research Institute; Andrew C Harris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center / Pediatric Stem Cell Transplantation and Cellular Therapies
Locations (16):
- United States (11):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Comprehensive Care Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - CHU Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schultz KR, Kariminia A, Ng B, Abdossamadi S, Lauener M, Nemecek ER, Wahlstrom JT, Kitko CL, Lewis VA, Schechter T, Jacobsohn DA, Harris AC, Pulsipher MA, Bittencourt H, Choi SW, Caywood EH, Kasow KA, Bhatia M, Oshrine BR, Flower A, Chaudhury S, Coulter D, Chewning JH, Joyce M, Savasan S, Pawlowska AB, Megason GC, Mitchell D, Cheerva AC, Lawitschka A, Azadpour S, Ostroumov E, Subrt P, Halevy A, Mostafavi S, Cuvelier GDE. Immune profile differences between chronic GVHD and late acute GVHD: results of the ABLE/PBMTC 1202 studies. Blood. 2020 Apr 9;135(15):1287-1298. doi: 10.1182/blood.2019003186. PMID 32047896
- [Background] Cuvelier GDE, Nemecek ER, Wahlstrom JT, Kitko CL, Lewis VA, Schechter T, Jacobsohn DA, Harris AC, Pulsipher MA, Bittencourt H, Choi SW, Caywood EH, Kasow KA, Bhatia M, Oshrine BR, Flower A, Chaudhury S, Coulter D, Chewning JH, Joyce M, Savasan S, Pawlowska AB, Megason GC, Mitchell D, Cheerva AC, Lawitschka A, West LJ, Pan B, Al Hamarneh YN, Halevy A, Schultz KR. Benefits and challenges with diagnosing chronic and late acute GVHD in children using the NIH consensus criteria. Blood. 2019 Jul 18;134(3):304-316. doi: 10.1182/blood.2019000216. Epub 2019 May 1. PMID 31043425